CLINICAL TRIAL: NCT05878717
Title: A Phase 2/3, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate The Efficacy And Safety of Belimumab Administered Subcutaneously in Adults With Systemic Sclerosis Associated Interstitial Lung Disease (SSC-ILD)
Brief Title: A Study of the Efficacy and Safety of Belimumab in Adults With Systemic Sclerosis Associated Interstitial Lung Disease
Acronym: BLISSc-ILD
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 218224; 2023-503219-14-01 (Registry Identifier: CTIS)
Record Dates: First submitted 2023-05-19; First posted 2023-05-26 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Systemic Sclerosis Associated Interstitial Lung Disease; Scleroderma, Systemic
Keywords: Monoclonal antibody; Autoimmune connective tissue disease; Skin; lung; systemic sclerosis; scleroderma; interstitial lung disease; belimumab
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse; Lung Diseases, Interstitial | interventions — belimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study where participant and investigator are masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Belimumab (Experimental): Participants will receive belimumab in addition to standard therapy.
  Interventions: Biological: Belimumab
- Placebo (Placebo Comparator): Participants will receive placebo in addition to standard therapy.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Belimumab — Belimumab will be administered.
  Other Names: BENLYSTA™, GSK1550188, LymphoStat-B™; BENLYSTATM, GSK1550188, LymphoStat-B™
  Arms: Belimumab
Other: Placebo — .Placebo will be administered.
  Arms: Placebo

SUMMARY:
This study investigates the efficacy and safety of belimumab compared to placebo, in addition to standard therapy, for the treatment of participants with systemic sclerosis associated interstitial lung disease (SSc-ILD). The study will evaluate the effect of belimumab treatment on lung function as well as on extra-pulmonary disease manifestations, including skin thickening and general symptoms, such as fatigue, that impact quality of life (QoL).

ELIGIBILITY:
Inclusion Criteria:

1. Participant is 18 years of age inclusive, or older at the time of signing the informed consent.
2. Documented diagnosis of SSc as defined by the American College of Rheumatology / European League Against Rheumatism 2013 SSc classification criteria.
3. Diffuse cutaneous disease, defined as presence of thickened skin with mRSS >0 over at least one skin area proximal to elbows and/or knees in addition to distal areas involvement on Day 1.
4. Total mRSS ≥15 on Day 1.
5. Evidence of interstitial lung disease on centrally read screening HRCT.
6. Anticentromere antibody negative on central test at screening.
7. Evidence for active or progressive disease
8. Participant has an area of uninvolved or mildly thickened skin that, in the opinion of the investigator, would allow SC injection at the abdomen or the front, middle region of the thigh.
9. Participant is capable and willing to self-administer the study medication or has a caregiver who is capable and willing to administer the study medication throughout the study.
10. A female participant is eligible to participate if she is not pregnant or breastfeeding, and one of the following conditions applies:

    Is a Woman of Non-Childbearing Potential (WONCBP) OR Is a Woman of Childbearing Potential (WOCBP) and using a contraceptive method that is highly effective.
11. Capable of giving signed informed consent.

Exclusion Criteria:

1. Systemic sclerosis-like illness, including but not limited to localized scleroderma (morphoea), eosinophilic fasciitis, sclerodermoid graft-versus-host disease, fibro mucinous conditions (scleroedema, scleromyxoedema), scleroderma-like conditions that are associated with environmental chemical and drug exposure (e.g., toxic rapeseed oil, vinyl chloride, bleomycin, gadolinium-based contrast agents [nephrogenic systemic fibrosis], or due to metabolic disease).
2. Primary diagnosis of a rheumatic autoimmune disease other than dcSSc, including but not limited to rheumatoid arthritis, systemic lupus erythematosus, polymyositis, dermatomyositis, systemic vasculitis, Sjogren's syndrome, antisynthetase syndrome, or mixed connective tissue disease, as determined by the investigator.
3. FVC ≤45% of predicted, or a DLco (corrected for hemoglobin) ≤40% of predicted or requiring supplemental oxygen at screening.
4. Pulmonary arterial hypertension, as determined by the investigator at, or prior to first day of dosing (Day 1).
5. SSc renal crisis within 6 months prior to the first day of dosing (Day 1).
6. History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematologic, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention or interfering with the interpretation of data.
7. Obstructive pulmonary disease (pre-bronchodilator FEV1/FVC <0.7).
8. Significant emphysema on screening HRCT (extent of emphysema exceeds extent of ILD).
9. Previous or planned major organ transplant (e.g., heart, lung, kidney, liver) or bone marrow transplant (e.g., autologous stem cell transplant).
10. Treatment with biologic agents, such as intravenous immunoglobulin or monoclonal antibodies, including marketed drugs, within 3 months or 5 half-lives (whichever is longer) prior to dosing.
11. Treatment with rituximab within 6 months prior to Day 1.
12. Treatment with non-biologic systemic immunosuppressive medication, other than mycophenolate, methotrexate or azathioprine (including, but not limited to cyclosporine A, tacrolimus, leflunomide, oral or parenteral gold, Janus kinase (JAK) inhibitors) within 3 months prior to Day 1.
13. Treatment with cyclophosphamide (oral or intravenous) within 6 months prior to Day 1.
14. Use of anti-fibrotic agents including colchicine, D-penicillamine, pirfenidone or tyrosine kinase inhibitors (e.g., nintedanib, nilotinib, imatinib, dasatinib) within 4 weeks prior to Day 1.
15. Cytotoxic drugs such as, chlorambucil, nitrogen mustard, or other alkylating agents within 6 months of Day 1.
16. Treatment with IM or IV corticosteroids within 1 month prior to Day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2029-05-17 (Estimated); Study Completion 2029-07-12 (Estimated)

PRIMARY OUTCOMES:
Absolute change from baseline in Forced Vital Capacity (FVC) millilitre (mL) at Week 52 | Baseline and Week 52

SECONDARY OUTCOMES:
Absolute change from baseline in modified Rodnan Skin Score (mRSS) at Week 52 | Baseline and Week 52
  The modified Rodnan Skin Score (mRSS) is an evaluation of the patients skin thickness rated by clinical palpation using a 0 to 3 scale. The scale differentiates between 0 = normal skin, 1 = mild thickness, 2 = moderate thickness, and 3 = severe thickness. The assessment is made across 17 pre-defined areas of the body, with total score ranging between 0 and 51. Higher scores indicate worse skin thickening.
Absolute change from baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue score at Week 52 | Baseline and Week 52
  FACIT-fatigue is a validated patient-reported measure developed originally to assess fatigue in individuals with cancer and has subsequently been used and validated in numerous chronic conditions, including SSc. FACIT-Fatigue scores range from 0-52 (higher scores indicate less fatigue).
Time to Systemic sclerosis (SSc) progression or death | From the date of assignment until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 52 Weeks
  SSc progression or death is defined as the time when major organ-based complications develop, or the participant dies.
Absolute change from baseline in FVC percentage (%) predicted at Week 52 | Baseline and Week 52
Relative decline from baseline in FVC (mL) greater than or equal to (≥)5% at Week 52 | Baseline and Week 52
Relative decline from baseline in FVC (mL) ≥10% at Week 52 | Baseline and Week 52
Absolute change from baseline in mRSS at Week 26 | Baseline and Week 26
  The modified Rodnan Skin Score (mRSS) is an evaluation of the patients skin thickness rated by clinical palpation using a 0 to 3 scale. The scale differentiates between 0 = normal skin, 1 = mild thickness, 2 = moderate thickness, and 3 = severe thickness with inability to pinch the skin into a fold. The assessment is made across 17 pre-defined areas of the body and therefore the total score can range from 0 to 51. Higher scores indicate worse skin thickening.
Proportion of participants achieving ≥20% increase in mRSS at Week 26 & 52 | At Week 26 and Week 52
Absolute change from baseline in Quantitative interstitial lung disease - whole lung (QILD-WL) at Week 52 | Baseline and Week 52
Absolute change from baseline in Quantitative lung fibrosis - whole lung (QLF-WL) at Week 52 | Baseline and Week 52
Proportion of participants achieving ≥2% increase in QILD at Week 52 | At Week 52
Absolute change from baseline in Carbon monoxide diffusing capacity (DLco) % predicted at Week 52 | Baseline and Week 52
Relative decline from baseline in DLco % predicted ≥15% at Week 52 | Baseline and Week 52
Absolute change from baseline in Cough Numeric Rating Scale (NRS) at Week 52 | Baseline and Week 52
  The cough NRS enables the participant to rate their cough on a defined scale from 0 to 10, where higher score indicating worse cough symptoms.
Absolute change from baseline in Scleroderma Skin Patient-Reported Outcome (SSPRO) at Week 52 | Baseline and Week 52
  SSPRO a patient-reported outcome (PRO) instrument developed to assess the skin-related quality of life (QoL) in participants with SSc. SSPRO has 18 items that assess four SSc skin-related HRQoL domain (emotional effects, physical effects, physical limitations and social effects). The higher score indicates worse impact on QoL.
Absolute change from baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) at Week 52 | Baseline and Week 52
  The HAQ-DI is a 26-question instrument assessing the degree of difficulty in accomplishing tasks in eight functional areas: dressing and grooming, arising, eating, walking, hygiene, reach, grip, and common daily activities. Each question is scored 0-3 (where 0=without difficulty & 3=unable to do). Higher scores reflect worse disability
Absolute change from baseline in Short Form-36 Health Survey Questionnaire (SF-36) at Week 52 | Baseline and Week 52
  The SF-36 yields an 8-scale profile of functional health and well-being scores as well as physical and mental component health summary scores. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
Absolute change from baseline in Patient Global Assessment of SSc Disease Activity (PtGA) at Week 52. | Baseline and Week 52
  PtGA is a patient reported outcome scale designed to capture the participants overall assessment of their disease. The participants are asked to score their disease on a scale from 0 to 10 where higher score indicates higher severity
Absolute change from baseline in Physician global assessment (PhGA) at Week 52 | Baseline and Week 52
  The PhGA is a score which enables the treating physician to rate the participants disease on a scale from 0 to 10, where higher score indicates greater severity.
Absolute change from baseline in Transition Dyspnea Index (TDI) at Week 52 | Baseline and Week 52
  TDI assess dyspnea severity over 3 components: functional impairment, magnitude of task and magnitude of effort. Each component has 7 grades, ranging from -3 (major deterioration) to +3 (major improvement), which are summed to calculate a score, ranging between -9 and +9. The lower the score the more severely the participant is affected by dyspnea.
Number of participants with Adverse Events (AEs), Adverse Events of special interest (AESIs) and Serious AEs (SAEs) up to Week 52 | Up to Week 52
Absolute change from baseline in DLco % predicted at Week 52 | Baseline and Week 52

CONTACTS AND LOCATIONS:
Locations (108):
- United States (20):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Upland, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, New Brunswick, New Jersey
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Potsdam, New York
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Denison, Texas
  - GSK Investigational Site, El Paso, Texas
  - GSK Investigational Site, Houston, Texas
- Argentina (3):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aire
- Australia (4):
  - GSK Investigational Site, Liverpool, New South Wales
  - GSK Investigational Site, Adelaide, South Australia
  - GSK Investigational Site, Woodville, South Australia
  - GSK Investigational Site, Fitzroy, Victoria
- Belgium (2):
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Liège
- Brazil (6):
  - GSK Investigational Site, Belo Horizonte
  - GSK Investigational Site, Curitiba
  - GSK Investigational Site, Juiz de Fora
  - GSK Investigational Site, Porto Alegre
  - GSK Investigational Site, Salvador
  - GSK Investigational Site, São Paulo
- China (11):
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Changchun
  - GSK Investigational Site, Chengdu
  - GSK Investigational Site, Luzhou
  - GSK Investigational Site, Mianyang
  - GSK Investigational Site, Nanjing
  - GSK Investigational Site, Nanning
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Shenyang
  - GSK Investigational Site, Xi'an
  - GSK Investigational Site, Zhuzhou
- Denmark (2):
  - GSK Investigational Site, Aarhus
  - GSK Investigational Site, Odense C
- GSK Investigational Site, Turku, Finland
- France (4):
  - GSK Investigational Site, Bobigny
  - GSK Investigational Site, Brest
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Toulouse
- Germany (5):
  - GSK Investigational Site, Cologne
  - GSK Investigational Site, Düsseldorf
  - GSK Investigational Site, Mainz
  - GSK Investigational Site, Minden
  - GSK Investigational Site, Tübingen
- Greece (4):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Heraklion Crete
  - GSK Investigational Site, Larissa
  - GSK Investigational Site, Thessaloniki
- Israel (6):
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Holon
  - GSK Investigational Site, Kfar Saba
  - GSK Investigational Site, Poria – Neve Oved
  - GSK Investigational Site, Ramat Gan
  - GSK Investigational Site, Tel Aviv
- Italy (14):
  - GSK Investigational Site, Ancona
  - GSK Investigational Site, Bari
  - GSK Investigational Site, Cagliari
  - GSK Investigational Site, Catania
  - GSK Investigational Site, Ferrara
  - GSK Investigational Site, Florence
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Modena
  - GSK Investigational Site, Napoli
  - GSK Investigational Site, Orbassano to
  - GSK Investigational Site, Padua
  - GSK Investigational Site, Pavia
  - GSK Investigational Site, Roma
  - GSK Investigational Site, Verona
- Japan (8):
  - GSK Investigational Site, Gunma
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokushima
  - GSK Investigational Site, Tokyo
- Mexico (4):
  - GSK Investigational Site, Chihuahua City
  - GSK Investigational Site, Guadalajara
  - GSK Investigational Site, Mérida
  - GSK Investigational Site, Torreón
- South Korea (2):
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon Kyunggi-do
- Spain (7):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Bilbao
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, VigoPontevedra
- United Kingdom (5):
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Leeds
  - GSK Investigational Site, London
  - GSK Investigational Site, Portsmouth
  - GSK Investigational Site, Wakefield

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/